CLINICAL TRIAL: NCT02531815
Title: A Randomized, Double-blind, Sponsor-open, Placebo-controlled, Single Intravenous Or Subcutaneous Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Pf-06741086 In Healthy Subjects And An Open-label Evaluation In Healthy Japanese Subjects
Brief Title: Dose Escalation Study of PF-06741086 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7841001; 2015-001821-17 (EudraCT Number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-25 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics; pharmacodynamics; Phase 1; first in human; monoclonal antibody; tissue factor pathway inhibitor; japanese
MeSH Terms: interventions — marstacimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1 (subcutaneous [SC]) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 2 (SC) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 3 (SC) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 4 (Intravenous [IV]) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 5 (IV) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 6 (IV) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 7 (IV) PF-06741086, Placebo (Experimental)
  Interventions: Biological: PF-06741086; Drug: Placebo
- Cohort 8 (subcutaneous [SC]) PF-06741086 (Experimental)
  Interventions: Biological: PF-06741086

INTERVENTIONS:
Biological: PF-06741086 — PF-06741086, single dose, beginning with Cohort 1 dose level at 30 mg. Subsequent dose levels will be determined after data review of prior cohort(s)
Drug: Placebo — Placebo for PF-06741086, single dose
  Other Names: saline placebo
  Arms: Cohort 1 (subcutaneous [SC]) PF-06741086, Placebo; Cohort 2 (SC) PF-06741086, Placebo; Cohort 3 (SC) PF-06741086, Placebo; Cohort 4 (Intravenous [IV]) PF-06741086, Placebo; Cohort 5 (IV) PF-06741086, Placebo; Cohort 6 (IV) PF-06741086, Placebo; Cohort 7 (IV) PF-06741086, Placebo

SUMMARY:
This Phase 1 first-in-human single ascending dose study will be a randomized, double-blind, placebo-controlled investigation of the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06741086.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs) and 100 kg (220 lbs).

Exclusion Criteria:

* Increased risk of thrombosis (coronary artery disease, hypercholesterolemia, diabetes)
* Use of nicotine/tobacco products
* Clotting disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs | Day 1 up to Day 84
Percentage of subjects with laboratory abnormalities | Day 1 up to Day 84
Number of subjects with change from baseline in vital signs | Day 1 up to Day 84
  blood pressure, pulse rate, temperature, respiration rate
Number of subjects with change from baseline in electrocardiogram (ECG) parameters | Day 1 to Day 84
Percentage of subjects with changes from baseline in physical examination | Day 1 to Day 84
Percentage of subjects with infusion site reactions | Day 1 up to Day 7
Percentage of subjects with injection site reactions | Day 1 to Day 7

SECONDARY OUTCOMES:
Plasma PF-06741086 concentrations | Day 1 up to Day 84
Maximum observed plasma concentration (Cmax) | Day 1 up to Day 84
Time for Cmax (Tmax) | Day 1 up to Day 84
Area under the curve from time zero to last quantifiable concentration (AUClast) | Day 1 up to Day 84
Terminal half-life (t 1/2) | Day 1 up to Day 84
Area under the plasma concentration-time profile from time zero extrapolated to infinite time (AUCinf) | Day 1 up to Day 84
Volume of distribution at steady state (Vss) | Day 1 up to Day 84
  Intravenous administration only
Apparent volume of distribution (Vz/F) | Day 1 up to Day 84
  Subcutaneous administration only
Clearance (CL) | Day 1 up to Day 84
  Intravenous administration only
Apparent clearance (CL/F) | Day 1 up to Day 84
  Subcutaneous administration only
Bioavailability (F) [F = AUC (inf,sc) / AUC (inf,iv)] | Day 1 up to Day 84
Mean residence time (MRT) | Day 1 up to Day 84
Total tissue factor pathway inhibitor concentrations over time | Day 1 up to Day 84
Thrombin generation | Day 1 up to Day 84
  may include lag time, peak thrombin generation, and endogenous thrombin generation potential
Prothrombin fragment 1+2 (PF1+2) concentrations over time | Day 1 up to Day 84
D-dimer concentrations over time | Day 1 up to Day 84
Dilute prothrombin time (dPT) | Day 1 up to Day 84
Frequency of anti-drug antibody (ADA) and neutralizing antibody (NAb) production | Day 1 up to Day 84
  Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7841001&StudyName=A%20Randomized%2C%20Double-blind%2C%20Sponsor-open%2C%20Placebo-controlled%2C%20Single%20Intravenous%20Or%20Subcutaneous%20Dose%20Escalation%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20Pf-06741086%20In%20Healthy%20Subjects%20And%20An%20Open-label%20Evaluation%20In%20Healthy%20Japanese%20Subjects